CLINICAL TRIAL: NCT02647606
Title: Comparison of the McGrath Videolaryngoscope and the Pentax-AWS With the Macintosh Laryngoscope for Nasotracheal Intubation in Patients With Manual In-line Stabilization
Brief Title: Comparison of the Videolaryngoscopes With Manual In-line Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, principal investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AJIRB-MED-DE1-15-334
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Oral Surgery; Maxillofacial Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- McGrath Group (Experimental): MgGrath videolaryngoscope will be used for nasotracheal intubation with MILS
  Interventions: Procedure: MILS; Device: McGrath videolaryngoscope
- Pentax-AWS Group (Experimental): Pentax-AWS videolaryngoscope will be used for nasotracheal intubation with MILS
  Interventions: Procedure: MILS; Device: Pentax AWS videolaryngoscope
- Macintosh Laryngoscope Group (Experimental): Macintosh Laryngoscope will be used for nasotracheal intubation with MILS
  Interventions: Procedure: MILS; Device: Macintosh laryngoscope

INTERVENTIONS:
Procedure: MILS — MILS(Manual in-line stabilization) will be applied during intubation. With MILS, different kinds of laryngoscope will be evaluated in a simulated difficult airway.
Device: McGrath videolaryngoscope — McGrath videolaryngoscope will be used for intubation
  Arms: McGrath Group
Device: Pentax AWS videolaryngoscope — Pentax AWS videolaryngoscope will be used for intubation
  Arms: Pentax-AWS Group
Device: Macintosh laryngoscope — Macintosh laryngoscope will be used for intubation
  Arms: Macintosh Laryngoscope Group

SUMMARY:
Videolaryngoscope is useful to improve the laryngeal view, especially during difficult intubation. There are several kinds of videolaryngoscopes and it is applicable during nasotracheal intubation. In this study, the investigators will compare the McGrath videolaryngoscope and Pentax-AWS with Macintosh laryngoscope for nasotracheal intubation in patients with manual in-line stabilization.

ELIGIBILITY:
Inclusion Criteria:

* oral or maxillofacial surgery
* ASA class I, II

Exclusion Criteria:

* anticipated difficult intubation
* necessity for rapid sequence induction
* cervical spine injury
* bleeding tendency

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
time for intubation | from holding the laryngoscope until the 1st ventilation after intubation, within 90 seconds
Cormack Lehane Laryngeal view | when laryngoscope is appropriately placed during intubation, approximately 2 seconds
POGP score | when laryngoscope is appropriately placed during intubation, approximately 2 seconds
  Percentage of glottic opening(POGO)

SECONDARY OUTCOMES:
external laryngeal manipulation | when laryngoscope is appropriately placed during intubation, approximately 2 seconds
  When the laryngeal view is insufficient during laryngoscope, another physician can manipulate the larynx externally to improve the laryngeal view. The necessity of external laryngeal manipulation will be recorded.
magill forceps | when laryngoscope is appropriately placed during intubation, approximately 5 seconds
  when the nasotracheal tube can not introduced to vocal cord manually, magill forceps can hold the tube to advance the tube through vocal cord. The necessity of magill forceps during intubation will be recorded
IDS (intubation difficulty scale) | during intubation, approximately 90 seconds
  IDS score is the sum of the following seven variables:
  N1: the number of intubation attempts>1 N2: the number of operators. 1 N3: the number of alternative intubation techniques used N4: glottic exposure (Cormack Lehane grade minus 1) N5: Lifting force required during laryngoscopy (0=normal; 1=increased) N6: necessity for external laryngeal pressure (0=not applied; 1=applied) N7: position of the vocal cords at intubation (0=abduction/ not visualized; 1=adduction)
numeric rating scale for intubation | during intubation, approximately 90 seconds
  0-10 (0; no difficulty, 10: hardest)
grade of bleeding | 10 seconds after completion of intubation
  After confirmation of successful intubation, Yankauer suction was introduced to access the intraoral bleeding during intubation.
  Grade is 4 points scale (none/trace/moderate/severe).

CONTACTS AND LOCATIONS:
Overall Officials: Go Un Roh, MD, Principal Investigator — Ajou University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roh GU, Kwak HJ, Lee KC, Lee SY, Kim JY. Randomized comparison of McGrath MAC videolaryngoscope, Pentax Airway Scope, and Macintosh direct laryngoscope for nasotracheal intubation in patients with manual in-line stabilization. Can J Anaesth. 2019 Oct;66(10):1213-1220. doi: 10.1007/s12630-019-01409-5. Epub 2019 May 29. PMID 31144258